CLINICAL TRIAL: NCT06718842
Title: Walking Program in Fatty Liver Children With Phenylketonuria: Response of Liver Enzymes
Brief Title: Walking Program in Fatty Liver Children With Phenylketonuria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, Department of Physical Therapy for Cardiovascular/Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005449
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Phenylketonurias; Non Alcoholic Fatty Liver
MeSH Terms: conditions — Phenylketonurias; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Experimental): this Group I will include PKU children sufferers (n=20) with non-alcoholic fatty liver that will perform walking program (online supervised free walking that will be applied daily for eight weeks)
  Interventions: Behavioral: walking free online supervised program
- Group II (No Intervention): this Group II will include PKU children sufferers (n=20) with non-alcoholic fatty liver that will act a waitlisted children

INTERVENTIONS:
Behavioral: walking free online supervised program — this Group I will include PKU children sufferers (n=20) with non-alcoholic fatty liver that will perform walking program (online supervised free walking that will be applied daily for eight weeks)
  Arms: group I

SUMMARY:
phenylketonuria (commonly known as PKU) is an inherited disorder that increases the levels of a substance called phenylalanine in the blood. PKU is usually associated with many metabolic complication including non-alcoholic fatty liver

DETAILED DESCRIPTION:
this study will include PKU children sufferers 9n=40) with non-alcoholic fatty liver to be randomly assigned to group I (n=20) that will perform walking program (online supervised free walking that will be applied daily for eight weeks) or group II (N=20) that will act as waitlisted children

ELIGIBILITY:
Inclusion Criteria:

* PKU children
* obese children
* fatty liver children (non-alcoholic fatty liver)

Exclusion Criteria:

* cardiac children
* diabetic children
* neurogenic disorders
* respiratory and renal problems

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — self-representation of gender identity
Enrollment: 40 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
alanine transamianse | it will be assessed after eight weeks
  it is a serum liver enzyme

SECONDARY OUTCOMES:
aspartate tranaminase | it will be assessed after eight weeks
  it is a serum liver enzyme
Gamma-glutamyl Transferase | it will be assessed after eight weeks
  it is a serum liver enzyme
alkaline phosphatase | it will be assessed after eight weeks
  it is a serum liver enzyme
triglycerides | it will be assessed after eight weeks
  it will be measured in the serum
body mass index | it will be assessed after eight weeks
  it will be measured after emptying bladder

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Study Chair — Cairo University
Locations (1):
- Cairo University, Dokki, Giza Governorate, Egypt